CLINICAL TRIAL: NCT03737682
Title: Hemostasis Achievement Reflecting Inflammatory Status of the Pulp Based on Cytokine Levels: A Cohort Study
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samah Mohsin, principal investigator, Cairo University
Other Study IDs: CEBD-CU-2018-10-31
Record Dates: First submitted 2018-10-31; First posted 2018-11-09 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hemostasis achievement: in which hemostasis at the exposure site was achieved in five minutes were included in group A
  Interventions: Diagnostic Test: ENzyme linked immunity-sorbet assays
- No hemostasis achievement: in which hemostasis at the exposure site couldn't be achieved in five minutes where included in group B
  Interventions: Diagnostic Test: ENzyme linked immunity-sorbet assays

INTERVENTIONS:
Diagnostic Test: ENzyme linked immunity-sorbet assays — Hemostasis achievement reflecting inflammatory status of the pulp based on cytokine levels

SUMMARY:
Assessment of pulp inflammation by hemostasis achievement after pulp exposure

DETAILED DESCRIPTION:
The possibility has been raised of diagnosing pulpal pathological status using the cytokines that are released during the inflammation process in healthy as well as infected tooth pulp. Cytokines are small polypeptides secreted by leucocytes and other inflammatory cells and are known to play important roles in the intensity and duration of the immune response

ELIGIBILITY:
Inclusion Criteria:

1. healthy children
2. patients had not used any inflammatory medications
3. primary molar teeth of these children were included based on the following clinical and radiographic criteria:

   1. no clinical symptoms or evidence of pulp degeneration (pain on percussion, history of swelling or sinus tract
   2. no spontaneous pain
   3. no radiographic signs of internal or external resorption, widened periodontal ligament space, or furcal/periapical radiolucency
   4. physiological root resorption of no more than one third the root length
   5. a deep caries lesion with a likelihood of pulp exposure during caries removal

Exclusion Criteria:

* patients used any anti-inflammatory medication

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: * primary teeth with carious pulp exposures during caries removal will be included in the study.
  * primary molars with the presence of exudate, purulence or necrotic pulp tissue around the exposure site will be excluded
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Measuring interleukin 2 (IL-2) | After 5 minutes
  to measure cytokines levels after coronal pulpal removal

SECONDARY OUTCOMES:
Measuring interleukin 6 (IL-6) and interleukin 8 (IL-8) | After 5 minutes
  to measure cytokines levels after coronal pulpal removal
Postoperative pain, Bifurcation/periapical radiolucency and Internal/external root resorption Or other pathological changes | 3,6,9,12 months
  To assess postoperative pain by verbal questioning and To observe presence or absence of radiolucency and root resorption or pathological condition

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt